CLINICAL TRIAL: NCT03880734
Title: Effects of Vitamin D3 Supplementation on Lung Functions and Exercise Tolerance in D3 Deficient Asthma COPD Overlap (ACO) Patients
Brief Title: This Study Include Asthma Chronic Obstructive Pulmonary Disease (COPD) Overlap Patients.Patients Were Vitamin D Deficient.Age Range 40-70 Years, Smokers.Patients Were Advised to Take Either Placebo or Vitamin D3.Lung Functions and Exercise Tolerance Were Assessed at Baseline and at 26th Weeks.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr.Naznin Sultana, principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10786
Record Dates: First submitted 2019-02-26; First posted 2019-03-19 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Asthma-COPD Overlap Syndrome
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: All the eligible patients were randomly assigned to either 'Study (A)' or 'Control (B)' group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): Vitamin D.Generic name-Cholecalciferol (40,000 IU).Dose- 80,000. Dosage-2 capsule/week for consecutive 26 weeks
  Interventions: Drug: Cholecalciferol
- control (Experimental): Placebo oral capsule.Dose 80,000.Dosage-2 capsules for consecutive 26 weeks
  Interventions: Other: Placebo oral capsule

INTERVENTIONS:
Drug: Cholecalciferol — ingredients-Cholecalciferol (40,000 IU),Microcrystalline Cellulose (58.1 gm),Butylated Hydroxy Toluene (0.2 mg),Magnesium Stearate (3 mg),Gelatin Capsule Shell (1 mg)
  Other Names: D-rise
  Arms: study
Other: Placebo oral capsule — ingredients- Microcrystalline Cellulose (303.8 gm),Butylated Hydroxy Toluene (0.2 mg),Magnesium Stearate (3 mg),Gelatin Capsule Shell (1 mg)
  Other Names: D-rise
  Arms: control

SUMMARY:
Vitamin D3 supplementation doen not change lung functions and exercise tolerance in vitamin D3 deficient ACO patient was the null hypothesis of the research.

DETAILED DESCRIPTION:
On the first day of enrollment, the objectives, nature, purpose and potential risk of all the procedures used for the study was explained in detail to each ACO patients (diagnosed by pulmonologist), with a cordial attitude giving emphasis on the benefits the participants might obtain from this study. The participants was encouraged for voluntary participation and was allowed to withdraw from the study even after participation, whenever participant felt uneasy. If the participant was agreed to be enrolled in the study, an informed written consent was taken in a prescribed form . Then all the patients were requested to attend the Department of Physiology at 8:30 am (after overnight fasting) on the examination day.

On that day, 10 ml of venous blood was collected from antecubital vein of patient in different vacutainer tubes and was taken to the laboratory of Department of Biochemistry and Molecular Biology as soon as possible, where 3 ml was for the estimation of serum vitamin D3 and rest was preserved at -4˚C.

If the patient was with D3 deficiency [Serum 25(OH)D <30 ng/ml], then the serum creatinine, serum HbA1C, serum parathormone (PTH), serum calcium (Ca2+), serum phosphate (PO43-), serum alkaline phosphatase (ALP), serum glutamate pyruvate transaminase (SGPT) serum cholesterol, serum High Density Lipoprotein (HDL), serum low density lipoprotein (LDL), serum triglyceride (TG), were assessed from the preserved blood. After getting all the biochemical reports the final selection was done, according to the inclusion and exclusion criteria.

Then all the eligible patients were randomly assigned to either 'Study (A)' or 'Control (B)' group.Then all the study variables of all the subjects of both the groups were assessed. These data were recorded as values of 'day 1' (A1, B1).

Subsequently a standard therapeutic treatment [according to Global Initiative for Chronic Obstructive Lung Diseases (GOLD) guideline] were prescribed (by the pulmonologist) to all the selected stable ACO patients of both groups. Proper education were given about drug, method of taking medication and medication plan plan, such as, training for Metered Dose Inhaler (MDI) use for 7 days.

Along with the standard pharmacological treatment of ACO, all patients of both the groups were advised to have sunlight exposure (within 11 am to 2 pm) only for 20 minutes daily and also to continue ad lib (according to their own choice) diet.

In addition, oral vitamin D3 (80,000 IU per week) and placebo were added to the treatment schedule of the 'Study' patients and 'Control' patients, respectively, for consecutive 13 weeks.

Subsequently, all these patients (of both groups) were cordially requested to attend the Department of Physiology on 13th week of their follow up, to reexamine all the study variables along with serum 25(OH)D and Ca (to check the toxicity or deficiency). Then according to serum level of 25(OH)D and Ca,[vitamin D3 40,000 IU (1 capsule) per one to six weeks] (American Vitamin D council 2018) was again given to the 'Study' patients for further 13 weeks. On the other hand, if serum 25(OH)D was <10 ng/ml [severely deficient (vitamin D Council 2018)] of any 'control' patient, then that participant was dropped out from the study (for ethical purpose) and a new ACO patient was enrolled to fulfil the desired sample number. After that they were cordially requested to visit again the Department of Physiology, BSMMU on '26th week' to reexamine all the study variables, and the data was recorded as values of '26th week' (A2, B2).

During the entire study period (26 weeks), a good rapport was kept by the researcher with every patient through taking time to time follow up over telephone and visiting patient's place with scheduled appointment to maintain a proper follow up at 2nd (at 13th week) and 3rd (at 26th week) visit of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonologist diagnosed patient of ACO
* Vitamin D3 deficient : Serum 25(OH)D <30 ng/ml
* Age: 40-70 years
* Sex: Male
* Socioeconomic status: middle class
* Smoker
* Anthropometric status:

BMI=18.6-24.9 kg mid upper arm circumference>25.1 cm waist-hip ratio<0.89

* Serum parathormone: 10-65 pg/ml
* Serum Ca2+: 8.5-10.5 mg/dl
* Serum PO43: 2.3-4.7 mg/dl
* Serum alkaline phosphatase: 30-120 U/L
* SGPT: <50 U/L
* Serum creatinine: 0.7-1.3 mg/dl
* Fasting Blood Sugar (FBS): 3.5-6.1 mmol/L
* Serum HbA1c: 4.5-6.3 %
* Serum cholesterol: <200 mg/dl
* Serum HDL: >40 mg/dl,
* Serum LDL: <130 mg/dl
* Serum TG: <150 mg/dl

Exclusion Criteria:

* With history of:

  * any other pulmonary diseases, as, chronic obstructive pulmonary disease bronchial asthma respiratory tract infection bronchiectasis pleural effusion tuberculosis interstitial lung disease pneumonectomy or pulmonary lobectomy
  * any cardiac disease, like - unstable angina pectoris congestive heart failure myocardial infarction cardiac arrhythmia
  * systemic hypertension
  * any liver disease
  * any malignancy
  * use of any drugs known to affect vitamin D metabolism within 1 month prior to study, as, antiepileptics (Phenytoin, Carbamazepine) antibiotics (Clotrimazole, Rifampicin) antihypertensives (Nifedipine, Spironolactone) antiretroviral drugs (Ritonavir, Saquinavir) endocrine drugs (Cyproterone acetate) glucocorticoids bisphosphonate calcium supplement
  * With biochemical evidence of diabetes mellitus renal insufficiency

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Lung function status measured by Forced vital capacity (FVC) | 8 month
  It is the volume of air that can be expired as forcefully and rapidly as possible after maximal inspiration.In adult male it is about 4.6 liters.
Lung function status measured by Forced expiratory volume in 1st second (FEV1) Mid Expiratory Flow 75% (MEF75%),Mid Expiratory Flow50% (MEF50%), Mid Expiratory Flow 25%(MEF25%) | 8 month
  When a person inspires maximally and exhales forcefully, then the volume, which is exhaled in 1st second is known as 'Forced Expiratory volume in 1st second'. It is normally 80% of forced vital capacity .
Lung function status measured by Ratio of Forced expiratory volume in 1st second and Forced vital capacity (FEV1 /FVC ratio) | 8 month
  It is the ratio of FEV1 to FVC expressed in percentage. FEV1/FVC ratio = FEV1/FVC×100. It is about 70% or higher.
Lung function status measured by Peak expiratory flow rate (PEER) | 8 month
  It is the maximum expiratory rate, beyond which the flow cannot be increased even with greatly increased additional force.
  In adult it is about 400-700 L/minute.
Forced Expiratory Flow25-75 (MEF25-75) | 8 month
  Forced expiratory flow during the middle half of the FVC.expressed in liters/second.
exercise tolerance measured by 6 Minute Walk Distancd (6MWD) | 8 month
  It is the distance that a person can quickly walk on a flat, hard surface in a period of 6 minutes.expressed in meters.
exercise tolerance measured by Oxygen saturation | 8 month
  Oxygen saturation is defined as the oxygen content expressed as a percentage
exercise tolerance measured by Level of dyspnea | 8 month
  a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity'.evaluated by BORG scale.
Exercise tolerance measured by level of fatigue | 8 month
  a subjective, unpleasant symptom which incorporates total body feelings ranging from tiredness to exhaustion, creating an unrelenting overall condition which interferes with individuals' .evaluated by BORG scale.

SECONDARY OUTCOMES:
Anthropomertric measurement measured by BMI | 8 month
  Body mass index (BMI) of each subject was calculated from the measured weight and height. Expressed in kg/m2
Anthropomertric measurement measured by mid upper arm circumference (MUAC) | 8 month
  measurement was done in cm
Anthropomertric measurement measured by waist hip ratio | 8 month
  Waist hip ratio was calculated as Weight in Cm/Height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Taskina Ali, MBBS, M.Phil, Study Director — Associate professor
Locations (1):
- BSMMU, Dhaka, Bangladesh

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03880734/Prot_SAP_ICF_000.pdf